CLINICAL TRIAL: NCT04857632
Title: Statin for Neuroprotection in Spontaneous Intracerebral Hemorrhage
Acronym: STATIC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STATIC
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Intracerebral Hemorrhage; Statins
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statins group (Experimental)
  Interventions: Drug: Statin
- Control group (No Intervention)

INTERVENTIONS:
Drug: Statin — atorvastatin 20mg per day for 7 days
  Arms: Statins group

SUMMARY:
Brain injury after spontaneous intracerebral hemorrhage results from pathophysiologic responses in the brain parenchyma due to hematoma formation, release of clot components, and surrounding edema. Inflammatory cascade activation in the perihematomal brain parenchyma has been implicated in the pathogenesis of secondary brain injury. Statins have been identified as a potential neuroprotective agent that targets the inflammatory response to intracerebral hemorrhage. In preclinical studies, statin treatment in animal intracerebral hemorrhage models has consistently demonstrated neuroprotective and recovery enhancement effects. Clinical investigations in humans reported better patient outcomes associated with statin use in patients with intracerebral hemorrhage, including reduced perihematomal edema, lower mortality rates, and improved functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* A clinical diagnosis of supratentorial intracerebral hemorrhage is confirmed by brain CT scan
* Hematoma volume ≤40ml
* The first dose of statin can be given within 24h of intracerebral hemorrhage symptom onset (if the patient is randomized to statin group)
* Written informed consent

Exclusion Criteria:

* Presence of intraventricular hemorrhage or subarachnoid hemorrhage
* Planned surgical hematoma evacuation by open craniotomy prior to randomization (planned minimally invasive surgery is not a contraindication to enrollment)
* Suspected secondary intracerebral hemorrhage related to trauma, tumor, ruptured aneurysm or arteriovenous malformation, hemorrhagic transformation of an ischemic infarct, Moyamoya disease, or venous sinus thrombosis
* Unable to swallow a statin pill and have contraindication to position a nasogastric tube
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST), or alanine aminotransferase (ALT) ≥2 × the upper limit of normal
* Known pregnancy, or positive pregnancy test, or breastfeeding
* Other diseases or abnormalities that the investigator believed might compromise the patient's safety during the study
* Historical modified Rankin scale score ≥2
* Life expectancy of less than 7 days
* Participation in another clinical study within 30 days prior to screening for the present study
* Prior use of statins within 1 month before intracerebral hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Age of 18 years or older
Enrollment: 98 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Perihemorrhagic edema to hematoma ratio | 7 days

SECONDARY OUTCOMES:
Absolute perihematomal edema changes | 7 days
Hematoma resolution rate | 7 days
Absolute hematoma volume changes | 7 days
Ordinal distribution of modified Rankin scale scores | 90 days
  The modified Rankin scale is a 7-point scale ranging from 0 (no symptoms) to 6 (death).
Proportion of patients with modified Rankin scale score 0-2 | 90 days
Proportion of patients with modified Rankin scale score 0-3 | 90 days
Rate of mortality | 30 dyas
National Institute of Health stroke scale | 7 days or discharge
  Scores on the National Institutes of Health Stroke Scale range from 0 to 42, with higher scores indicating more severe neurologic deficits.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Fengtai Youanmen Hospital, Beijing, Beijing Municipality
  - Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Hebei Province Shunping County Hospital, Baoding

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gao D, Chu X, Zhang Y, Yan H, Niu L, Jiang X, Bao S, Ji X, Wu C. Statins for neuroprotection in spontaneous intracerebral haemorrhage (STATIC): protocol for a multicentre, prospective and randomised controlled trial. BMJ Open. 2024 Jun 21;14(6):e079879. doi: 10.1136/bmjopen-2023-079879. PMID 38908848